CLINICAL TRIAL: NCT07082140
Title: The Effect of Social Media-Based Education on the Knowledge and Attitudes of Women of Childbearing Age in the Preconception Period and on Healthy Lifestyle Behaviors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBU-AYDINKARTAL-012
Record Dates: First submitted 2024-12-07; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Social Media Based Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (n:40) (Experimental): Participants in the intervention group will be required to follow the Instagram account created specifically for the training. The Instagram account will be made private to prevent women in the control group from accessing Instagram posts. The training provided via Instagram will last 2 weeks, including the process of sharing all posts and videos. After the completion of the training, the "Healthy Lifestyle Behaviors Scale" and the "Preconceptional Knowledge and Attitude Scale" will be applied as a post-test.
  Interventions: Other: Social media based education
- Control group (n:40 (No Intervention): No application will be made. After all stages of the research are completed, training will be applied to the control group participants. After the research is completed, all participants will be given a brochure containing the information in the training content.

INTERVENTIONS:
Other: Social media based education — Participants in the intervention group will be required to follow the Instagram account created specifically for the training. The Instagram account will be made private to prevent women in the control group from accessing Instagram posts. The training provided via Instagram will last 2 weeks, including the process of sharing all posts and videos. After the completion of the training, the "Healthy Lifestyle Behaviors Scale" and the "Preconceptional Knowledge and Attitude Scale" will be applied as a post-test.
  Arms: Intervention group (n:40)

SUMMARY:
In order to determine the effect of education provided through social media on the knowledge and attitudes of women of childbearing age during the preconceptional period and its relationship with healthy lifestyle behaviors, a randomized controlled pre-test and post-test design and control group was planned. The research universe will consist of women of childbearing age who applied to Ümraniye Education and Research Hospital, agreed to participate in the study and met the inclusion criteria (N: 80). In this randomized controlled pre-test and post-test design and control group study, in order to determine the sample size; the data were normally distributed, the standard deviation of the main mass was estimated as 1 and the effect size (difference) was estimated as 0.8. For the analysis to be conducted, it was calculated that the highest power value of the study would be 0.942182 if two independent n₁=40, n₂=40 samples were taken at a significance level of 5%. The G-power analysis result is given below. In addition, after the data collection, the adequacy of the sample size in the study will be evaluated with a post hoc power analysis. Women who volunteer to participate in the study will be assigned to the intervention and control groups using a computer-aided simple random sampling method. Computer-aided randomization will be used in the study, and the number of cases will be entered through the program with the URL address https://www.randomizer.org and random assignment will be made to the intervention and control groups. Preconceptional period education will be provided to the women in the intervention group via social media. No application will be made to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being willing to participate in the study.
* Being a woman of childbearing age
* Planning to get pregnant within 1 year
* Using Instagram and WhatsApp

Exclusion Criteria:

- Being pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-05 (Estimated); Primary Completion 2025-12-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 10 minutes
  This form, created by researchers based on literature, includes questions about the participants' age, obstetric history, healthy lifestyle behaviors, etc.
Healthy Lifestyle Behaviors Scale (HLBS-II) | 10 minutes
  The scale, whose validity and reliability study was conducted in our country by Bahar et al. in 2008, was developed by Walker et al. in 1996 to measure the health-enhancing behaviors of the individual in relation to a healthy lifestyle. The scale has six sub-dimensions: health responsibility (3,9,15,21,27,33,39,45,51), physical activity (4,10,16,22,28,34,40,46), nutrition (2,8,14,20,26,32,38,44,50), spiritual development (6,12,18,24,30,36,42,48,52), interpersonal relations (1,7,13,19,25,31,37,43,49) and stress management (5,11,17,23,29,35,41,47) and consists of a total of 52 items. The interpersonal relations scale sub-dimension evaluates the relationships between the individual and the environment. Communication is necessary in a healthy relationship.
Preconceptional Knowledge and Attitude Scale | 10 minutes
  It was developed by Gökdemir and Eryılmaz in 2022. The original language of the scale is Turkish and it is a 5-point Likert type. The scale can be applied to married and single women between the ages of 18-45 who are of childbearing age. The Preconceptional Knowledge and Attitude Scale consists of a total of 43 items, 42 positive (straight) and 1 negative (reverse) item, and 7 sub-dimensions (factors). The distribution of the items in the scale to the factors is as follows. Factor 1 (Attitudes Towards Preconceptional Health Protection and Development): There are a total of 10 items in this dimension, consisting of items 10, 15, 17, 18, 19, 21, 23, 25, 26, and 31. Factor 2 (Attitudes Towards Fertility Planning): This dimension consists of items 28, 30, 32, 34, 38, 39, and 40, and has a total of 7 items. Factor 3 (Attitudes Towards Living Conditions Before Having Children): This dimension consists of items 27, 29, 41, 35, and 42, and has a total of 5 items.

SECONDARY OUTCOMES:
Introductory Information Form | 10 minutes
  This form, created by researchers based on literature, includes questions about the participants' age, obstetric history, healthy lifestyle behaviors, etc.
Healthy Lifestyle Behaviors Scale (HLBS-II) | 10 minutes
  The scale, whose validity and reliability study was conducted in our country by Bahar et al. in 2008, was developed by Walker et al. in 1996 to measure the health-enhancing behaviors of the individual in relation to a healthy lifestyle. The scale has six sub-dimensions: health responsibility (3,9,15,21,27,33,39,45,51), physical activity (4,10,16,22,28,34,40,46), nutrition (2,8,14,20,26,32,38,44,50), spiritual development (6,12,18,24,30,36,42,48,52), interpersonal relations (1,7,13,19,25,31,37,43,49) and stress management (5,11,17,23,29,35,41,47) and consists of a total of 52 items. The interpersonal relations scale sub-dimension evaluates the relationships between the individual and the environment. Communication is necessary in a healthy relationship.
Preconceptional Knowledge and Attitude Scale | 10 minutes
  It was developed by Gökdemir and Eryılmaz in 2022. The original language of the scale is Turkish and it is a 5-point Likert type. The scale can be applied to married and single women between the ages of 18-45 who are of childbearing age. The Preconceptional Knowledge and Attitude Scale consists of a total of 43 items, 42 positive (straight) and 1 negative (reverse) item, and 7 sub-dimensions (factors). The distribution of the items in the scale to the factors is as follows. Factor 1 (Attitudes Towards Preconceptional Health Protection and Development): There are a total of 10 items in this dimension, consisting of items 10, 15, 17, 18, 19, 21, 23, 25, 26, and 31. Factor 2 (Attitudes Towards Fertility Planning): This dimension consists of items 28, 30, 32, 34, 38, 39, and 40, and has a total of 7 items. Factor 3 (Attitudes Towards Living Conditions Before Having Children): This dimension consists of items 27, 29, 41, 35, and 42, and has a total of 5 items.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No